CLINICAL TRIAL: NCT00186654
Title: Acupuncture and Massage for Depression During Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HS09988
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture
Procedure: Perinatal massage

SUMMARY:
This study evaluates the efficacy of acupuncture and massage for the treatment of depression during pregnancy. The study also examines differential effects of study treatments on delivery outcome and post partum depression.

DETAILED DESCRIPTION:
Participants in this study are randomly assigned to one of the three experimental groups that include two types of acupuncture treatment and perinatal massage. The two acupuncture treatments are delivered in a double-blind fashion. Treatments consist of an acute phase during which participants receive 12 treatment sessions over a period of 8 weeks. Responders and partial responders enter a continuation phase during which they receive weekly treatments that end 10 weeks post delivery. At the end of the continuation phase, participants continue to be clinically assessed at 3 and 6 months after the end of treatment to detail the natural course of relapse to the index episode in the three treatment groups.

ELIGIBILITY:
Inclusion Criteria:- Meet criteria for a current major depressive episode with an HRSD(17) score of at least 14.

* Ambulatory women (age³18) with a viable pregnancy,
* Pregnancy between 22 and 30 weeks of gestation
* Fluent in English

Exclusion Criteria:- Meeting criteria for a primary Axis I disorder in past 2 months, other than unipolar depression or social phobia

* Seasonal affective disorder or episode duration of 2 years or more (chronic depression)
* Abnormal results on a laboratory screen that will include a thyroid panel and a drug screen.
* Serious uncontrolled medical conditions or conditions that may be a medical basis of a depression.
* Cluster B personality disorders.
* Confounding treatments for depression, including any psychotherapy, herbs, or pharmacotherapy.
* Current use of any prescribed psychotropic medication or any medication that impacts mood.
* Treatment with ECT or vagal nerve stimulation during the last year.
* Current active suicidal potential necessitating immediate treatment.
* Absence of prenatal care from an OBGYN practitioner in the community.
* Any condition that necessitates bed rest.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180

PRIMARY OUTCOMES:
Depression severity and response status after 8 weeks of treatment

SECONDARY OUTCOMES:
Depression severity at 3, 6, & 9 months post partum; delivery outcome

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Manber, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Manber R, Schnyer RN, Lyell D, Chambers AS, Caughey AB, Druzin M, Carlyle E, Celio C, Gress JL, Huang MI, Kalista T, Martin-Okada R, Allen JJB. Acupuncture for depression during pregnancy: a randomized controlled trial. Obstet Gynecol. 2010 Mar;115(3):511-520. doi: 10.1097/AOG.0b013e3181cc0816. PMID 20177281